CLINICAL TRIAL: NCT02585921
Title: Combining, Expanding, and Evaluating Multiple Evidence-based Organ Donation Interventions
Brief Title: Organ Donation Interventions Among High Students
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment completed.
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Daryl Thornton, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1 R39OT26989-01-00; R39OT26989- (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Tissue and Organ Procurement; Adolescent Behavior; Communication
Keywords: Urban Health
MeSH Terms: conditions — Adolescent Behavior; Communication

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Health & Wellness (No Intervention): Following enrollment, participants will learn about health and wellness.
- Organ Donation Video Education (Experimental): Following recruitment, participants will watch and discuss videos about organ donation.
  Interventions: Behavioral: Video Interventions
- Organ Donation Discussion Education (Experimental): Following recruitment, participants will learn techniques to introduce and discuss the topic of organ donation with parents or guardians.
  Interventions: Behavioral: Donation Discussion Education
- Both Video and Discussion Education (Experimental): Following recruitment, participants will watch and discuss videos about organ donation and then learn techniques to introduce and discuss the topic of organ donation with parents and guardians.
  Interventions: Behavioral: Video Interventions; Behavioral: Donation Discussion Education

INTERVENTIONS:
Behavioral: Video Interventions — Participants will watch 2 5-minute videos and then discuss them as a group.
  Arms: Both Video and Discussion Education; Organ Donation Video Education
Behavioral: Donation Discussion Education — Participants will learn techniques for introducing and discussing organ donation with parents and guardians.
  Arms: Both Video and Discussion Education; Organ Donation Discussion Education

SUMMARY:
The number of persons actively waiting on the national solid organ waiting list continues to rise while the number donating organs has failed to keep pace. This is a particular problem for some portions of northeastern Ohio where the donation rate is as low as 32%. Adolescents are an important group for organ donation efforts as they have not yet applied for a driver's license and represent the majority of future donors. Yet many organ donation interventions have not targeted adolescents. The investigators propose to utilize existing high school teen summits developed by our Consortium partners to evaluate the effectiveness of existing donation interventions. Together, the investigators will conduct a randomized controlled 2x2 factorial trial to evaluate the independent and combined effects of two donor education interventions on consent for organ donation on the electronic Ohio Donor Registry. One thousand six hundred students over the age of 15.5 years from Cleveland-area high schools will be enrolled.

DETAILED DESCRIPTION:
Over 74,000 people are actively waiting for a solid organ to improve and extend their lives yet each year the number of deceased donors remains less than 11,000.1 Substantial changes are needed to increase the number of donated organs or many persons in need of a transplant will die without receiving one. The major limiting factor to organ donation remains the low consent rate.2 Increasing consent for organ donation will likely increase both the availability of organs and, by extension, increase the duration and quality of life of those waiting.3,4 While most people who consent to organ donation do so while obtaining their driver's licenses at the bureau of motor vehicles,5,6 the bureau of motor vehicles' staff generally do not have the training to provide sufficient information to answer questions regarding donation. As a result, bureau of motor vehicle patrons may not be receiving the information necessary to allay their fears and concerns sufficiently enough to provide informed consent for donation. We have previously demonstrated that adolescents have concerns regarding organ donation that stem from lack of knowledge about the process and from a paucity of discussions regarding organ donation with their parents.7 We and others have also found that efforts to increase consent for organ donation among adolescents must address altruism regarding donation and the positive effects of donation.8,9. We incorporated these findings into the development of a video intervention tailored towards adolescents. In a community-based randomized trial, we found that the video was effective in increasing consent for organ donation.10 This project incorporated the successful aspects of these multiple organ donation interventions to facilitate consent for organ donation among adolescents.

Our consortium partners, the Cleveland branch of the Minority Organ and Tissue Transplant Education Program (Cleveland MOTTEP), Lifebanc (the Organ Procurement Organization for Northeast Ohio), the Cleveland Eye Bank, and the Kidney Foundation of Ohio, had been collaborating to conduct twice yearly organ donation summits for adolescents for almost 10 years. The summits were 1-day meetings of 100 - 150 students from 5 high schools in Cleveland and the surrounding neighborhoods. The goals of the summits were to increase knowledge and awareness of organ and tissue donation and transplantation, as well as to assist in chronic disease prevention. While the summits have become a mainstay in the community, they have been limited in scope, devoid of a uniform curriculum, variable in execution, and have lacked formal evaluation.

The purpose of this study was to expand on the existing high school education summits by creating and implementing a uniform, validated organ donation curriculum based on successful best practices with integration of successful organ donation video interventions and by rigorously evaluating the effect of the individual and combined components. We employed a 2x2 factorial randomized design to explore the independent and combined effects of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Not previously consented to organ donation
* Attending high school or GED-granting school

Exclusion Criteria:

* Non-English speaking
* Visually impaired
* Cognitively impaired

Ages: 15 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 872 (Actual)
Dates: Start 2015-10; Primary Completion 2017-05-31 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who consent to donate organs | 1 month
  Consent on the electronic donor registry

SECONDARY OUTCOMES:
Proportion of participants who reported having donation discussions with their parents | 1 month
  Proportion of participants who reported having donation discussions with their parents
Proportion of participants' parents who consent to donate organs | 1 month
  Proportion of participants' parents who consent to donate organs

CONTACTS AND LOCATIONS:
Overall Officials: John D Thornton, MD, MPH, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States